CLINICAL TRIAL: NCT07380893
Title: Prevalence of Left Ventricular Hypertrophy (LVH) in CKD Patients and Effect of Erythropoietin Therapy
Brief Title: Left Ventricular Hypertrophy in CKD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Mohamedin, resident of internal medicine, Sohag University
Other Study IDs: Soh-Med--25-11-7MS
Record Dates: First submitted 2025-12-30; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: transthoracic echocardiography — Standard transthoracic echocardiography will be performed for all participants, measuring:
  * Left ventricular end-diastolic diameter (LVEDD)
  * Interventricular septal thickness (IVSD)
  * Posterior wall thickness (PWD)
  * Left ventricular mass (LVM)
  * Left ventricular mass index (LVMI = LVM/body surface area)

SUMMARY:
The goal of this observational study is to determine the prevalence of left ventricular hypertrophy among patients with chronic kidney disease at Sohag University Hospital and assess the effect of erythropoietin therapy on left ventricular mass and geometry in anemic CKD patients.

The main question it aims to answer is:

Does erythropoietin therapy mitigate or even reverse LVH and improve cardiac geometry ?

DETAILED DESCRIPTION:
The prevalence of LVH in CKD patients has been reported to range from 40% to 75%, depending on disease stage, blood pressure control, and diagnostic methodology. LVH typically develops early and worsens with CKD progression, reflecting the close interplay between renal dysfunction and cardiac remodeling.

Anemia is a prominent non-hemodynamic contributor to LVH in CKD. Reduced erythropoietin (EPO) production by the damaged kidneys, together with iron deficiency and chronic inflammation, leads to decreased oxygen delivery, compensatory cardiac output elevation, and subsequent ventricular hypertrophy.

Given the strong association between CKD, anemia, and cardiovascular remodeling, investigating the prevalence of LVH and the effect of erythropoietin therapy on left ventricular mass among CKD patients can provide critical insights into optimizing cardiovascular risk management in this high-risk group.

this study will be conducted to :

1. To determine the prevalence of left ventricular hypertrophy among patients with chronic kidney disease at Sohag University Hospital.
2. To assess the effect of erythropoietin therapy on left ventricular mass and geometry in anemic CKD patients.

A total of 100 CKD patients will be included.

* Phase I : All CKD patients will undergo echocardiographic evaluation to determine the prevalence of LVH.
* Phase II : Among anemic CKD patients with LVH receiving erythropoietin therapy , will be followed for 6 months

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with CKD stages 3-5.
* Stable clinical condition for ≥3 months.
* Anemia (Hb <10 g/dL) for cohort phase.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Valvular or ischemic heart disease.
* Uncontrolled hypertension (BP >180/110 mmHg).
* Acute coronary syndrome or decompensated heart failure in the past 3 months.
* Malignancy or active infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study population is adults age (18-75)years, diagnosed with CKD stage 3-5 .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in LVMI following erythropoietin therapy in anemic CKD patients. | - baseline transthoracic echocardiography will be performed for all group study.

SECONDARY OUTCOMES:
Association between hemoglobin level and LVMI. | 6 months of erythropoitin therapy , transthoracic echocardiography will be performed for all group study.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Kh Ahmed, MD, Study Chair — Sohag university- faculty of medicine - internal medicine department